CLINICAL TRIAL: NCT01162889
Title: Ascending Single Dose Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of ATR-107 Administered Subcutaneously And Intravenously To Healthy Subjects
Brief Title: Study To Assess The Safety And Tolerability Of Increasing Single Doses Of ATR-107 (PF-05230900) In Healthy People
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B2281001; 3243K1-1000
Record Dates: First submitted 2010-06-09; First posted 2010-07-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: pharmacokinetics; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — ATR-107; Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Placebo - SC injection (Placebo Comparator)
  Interventions: Drug: Placebo SC Injection
- Drug dose level 1 - SC injection (Experimental)
  Interventions: Drug: ATR-107 (PF-05230900) SC Injection
- Drug dose level 2 - SC injection (Experimental)
  Interventions: Drug: ATR-107 (PF-05230900) SC Injection
- Drug dose level 3- SC injection (Experimental)
  Interventions: Drug: ATR-107 (PF-05230900) SC Injection
- Drug dose level 4 - SC injection (Experimental)
  Interventions: Drug: ATR-107 (PF-05230900) SC Injection
- Drug dose level 5 - SC injection (Experimental)
  Interventions: Drug: ATR-107 (PF-05230900) SC Injection
- Drug dose level 6 - IV Infusion (Experimental)
  Interventions: Drug: ATR-107 (PF-05230900) IV Infusion
- Drug dose level 7 - IV Infusion (Experimental)
  Interventions: Drug: ATR-107 (PF-05230900) IV Infusion
- Drug dose level 8 - IV infusion (Experimental)
  Interventions: Drug: ATR-107 (PF-05230900) IV Infusion
- Placebo - IV infusion (Placebo Comparator)
  Interventions: Drug: Placebo IV Infusion
- Drug dose level 9 - IV infusion (Experimental)
  Interventions: Drug: ATR-107 (PF-05230900) IV Infusion

INTERVENTIONS:
Drug: Placebo SC Injection — Single injection
  Arms: Placebo - SC injection
Drug: ATR-107 (PF-05230900) SC Injection — Single intravenous infusion, 60 minute duration
  Arms: Drug dose level 1 - SC injection
Drug: ATR-107 (PF-05230900) SC Injection — Single subcutaneous injection
  Arms: Drug dose level 2 - SC injection
Drug: ATR-107 (PF-05230900) SC Injection — Single subcutaneous injection
  Arms: Drug dose level 3- SC injection
Drug: ATR-107 (PF-05230900) SC Injection — Single subcutaneous injection
  Arms: Drug dose level 4 - SC injection
Drug: ATR-107 (PF-05230900) SC Injection — Single subcutaneous injection
  Arms: Drug dose level 5 - SC injection
Drug: ATR-107 (PF-05230900) IV Infusion — Single subcutaneous injection
  Arms: Drug dose level 6 - IV Infusion
Drug: ATR-107 (PF-05230900) IV Infusion — Single intravenous infusion, 60 minute duration
  Arms: Drug dose level 7 - IV Infusion
Drug: ATR-107 (PF-05230900) IV Infusion — Single intravenous infusion, 60 minute duration
  Arms: Drug dose level 8 - IV infusion
Drug: Placebo IV Infusion — Single intravenous infusion, 60 minute duration
  Arms: Placebo - IV infusion
Drug: ATR-107 (PF-05230900) IV Infusion — Single intravenous infusion, 60 minute duration
  Arms: Drug dose level 9 - IV infusion

SUMMARY:
This is a "first in human" study to determine the safety and tolerability of the drug after single doses. Nine doses of increasing strength will be injected or infused (given into a vein) to 9 different groups of people. One third of the participants will be given an injection or infusion of placebo (sugar water). All participants will be healthy people.

DETAILED DESCRIPTION:
First in human single dose study. Study terminated 12 October 2011. The ATR-107 Development team reached a recommendation to terminate further development of ATR-107 (PF-05230900). This was based on a number of factors, including development of anti-drug antibodies in approximately 70% of subjects in the First-in-Human study in healthy volunteers (B2281001). This recommendation is not based on adverse events observed in study B2281001.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential
* Body mass index between 17.5 to 30.5 and body weight > 50 kg

Exclusion Criteria:

* History of significant medical illness
* Positive urine drug screen or alcohol dependance
* Smoking > 10 cigarettes per day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent AEs and SAEs, AEs leading to withdrawal, immunogenicity, injection and infusion reactions, and clinically significant changes in laboratory tests, vital signs and ECGs if reported. | 20 months
Pharmacokinetics parameters - Cmax, Tmax, AUC(0-oo), AUClast, t 1/2, CL and Vz | 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Overland Park, Kansas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2281001&StudyName=Study%20To%20Assess%20The%20Safety%20And%20Tolerability%20Of%20Increasing%20Single%20Doses%20Of%20ATR-107%20%28PF-05230900%29%20In%20Healthy%20People